CLINICAL TRIAL: NCT02380313
Title: A Phase I, Open-Label, Dose-Finding Study of Afuresertib Administered in Combination With Either Enzalutamide (Xtandi) or Abiraterone (Zytiga) in Male Subjects With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Dose-Finding Study of Afuresertib Administered in Combination With Either Enzalutamide or Aibraterone
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study cancelled: Withdrawn before enrollment of any participants
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201672
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Cancer
Keywords: Metastatic Castration-Resistant Prostate Cancer; Enzalutamide; Abiraterone; Dose-Finding; Afuresertib
MeSH Terms: conditions — Neoplasms | interventions — afuresertib; enzalutamide; abiraterone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Afuresertib 125 mg + enzalutamide 160 mg (Experimental): Participants will be receiving enzalutamide at the recommended dose for at least 4 weeks prior to enrolment into this cohort. Afuresertib 125mg and enzalutamide 160 mg will be dosed continuously on a once daily schedule for 28-day intervals.
  Interventions: Drug: Afuresertib; Drug: Enzalutamide
- Afuresertib 150 mg + enzalutamide 160 mg (Experimental): Participants will be receiving enzalutamide at the recommended dose for at least 4 weeks prior to enrolment into this cohort. Afuresertib 150 mg and enzalutamide 160 mg will be dosed continuously on a once daily schedule for 28-day intervals.
  Interventions: Drug: Afuresertib; Drug: Enzalutamide
- Afuresertib 175 mg + enzalutamide 160 mg (Experimental): Participants will be receiving enzalutamide at the recommended dose for at least 4 weeks prior to enrolment into this cohort. Afuresertib 175 mg and enzalutamide 160 mg will be dosed continuously on a once daily schedule for 28-day intervals.
  Interventions: Drug: Afuresertib; Drug: Enzalutamide
- Afuresertib 200 mg + enzalutamide 160 mg (Experimental): Participants will be receiving enzalutamide at the recommended dose for at least 4 weeks prior to enrolment into this cohort. Afuresertib 200 mg and enzalutamide 160 mg will be dosed continuously on a once daily schedule for 28-day intervals.
  Interventions: Drug: Afuresertib; Drug: Enzalutamide
- Afuresertib 125 mg + abiraterone 1000 mg + prednisone 5 mg (Experimental): Participants will be receiving abiraterone at the recommended dose for at least 2 weeks prior to enrolment into this cohort. Afuresertib 125mg and abiraterone 1000 mg will be dosed continuously on a once daily schedule for 28-day intervals. Continuous BID prednisone 5mg will be coadministered per the labelled recommendations.
  Interventions: Drug: Afuresertib; Drug: Abiraterone; Drug: Prednisone
- Afuresertib 150 mg + abiraterone 1000 mg + prednisone 5 mg (Experimental): Participants will be receiving abiraterone at the recommended dose for at least 2 weeks prior to enrolment into this cohort. Afuresertib 150mg and abiraterone 1000 mg will be dosed continuously on a once daily schedule for 28-day intervals. Continuous BID prednisone 5mg will be coadministered per the labelled recommendations.
  Interventions: Drug: Afuresertib; Drug: Abiraterone; Drug: Prednisone
- Afuresertib 100 mg + abiraterone 1000 mg + prednisone 5 mg (Experimental): Participants will be receiving abiraterone at the recommended dose for at least 2 weeks prior to enrolment into this cohort. Afuresertib 100 mg and abiraterone 1000 mg will be dosed continuously on a once daily schedule for 28-day intervals. Continuous BID prednisone 5mg will be coadministered per the labelled recommendations.
  Interventions: Drug: Afuresertib; Drug: Abiraterone; Drug: Prednisone
- RP2D of Afuresertib + enzalutamide 160 mg (Experimental): Participants in this arm will receive RP2D of afuresertib established in escalation cohort in addition to plus enzalutamide 160 mg once daily.
  Interventions: Drug: Afuresertib; Drug: Enzalutamide
- Afuresertib RP2D + abiraterone 1000 mg + prednisone 5 mg (Experimental): Participants in this arm will receive RP2D of afuresertib established in escalation cohort in addition to abiraterone 1000 mg once daily and continuous BID prednisone 5 mg coadministered per the labelled recommendations.
  Interventions: Drug: Afuresertib; Drug: Abiraterone; Drug: Prednisone
- Afuresertib RP2D + abiraterone + prednisone in PK cohort (Experimental): Participants in this arm will receive RP2D of afuresertib established in escalation cohort in addition to abiraterone 1000 mg once daily and continuous BID prednisone 5 mg coadministered per the labelled recommendations
  Interventions: Drug: Afuresertib; Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: Afuresertib — White of off-white round immediate release tablet for oral administration with unit dose strength of 50 mg and 75 mg to achieve the dosage level of 100 mg, 125 mg, 150 mg or 200 mg once daily.
Drug: Enzalutamide — Opaque white to off-white capsule for oral administration with unit dose strength of 40mg to achieve dose level of 160 mg once daily.
  Arms: Afuresertib 125 mg + enzalutamide 160 mg; Afuresertib 150 mg + enzalutamide 160 mg; Afuresertib 175 mg + enzalutamide 160 mg; Afuresertib 200 mg + enzalutamide 160 mg; RP2D of Afuresertib + enzalutamide 160 mg
Drug: Abiraterone — White to off-white tablet for oral administration with unit dose strength 250 mg to achieve dose level of 1000 mg once daily.
  Arms: Afuresertib 100 mg + abiraterone 1000 mg + prednisone 5 mg; Afuresertib 125 mg + abiraterone 1000 mg + prednisone 5 mg; Afuresertib 150 mg + abiraterone 1000 mg + prednisone 5 mg; Afuresertib RP2D + abiraterone + prednisone in PK cohort; Afuresertib RP2D + abiraterone 1000 mg + prednisone 5 mg
Drug: Prednisone — Continuous twice daily co administration of prednisone 5 mg as per labelled recommendation from United State Prescribing Information.
  Arms: Afuresertib 100 mg + abiraterone 1000 mg + prednisone 5 mg; Afuresertib 125 mg + abiraterone 1000 mg + prednisone 5 mg; Afuresertib 150 mg + abiraterone 1000 mg + prednisone 5 mg; Afuresertib RP2D + abiraterone + prednisone in PK cohort; Afuresertib RP2D + abiraterone 1000 mg + prednisone 5 mg

SUMMARY:
This study is being conducted to characterize the safety and recommended phase 2 dose (RP2D) of combining afuresertib, independently with 2 approved drugs: enzalutamide (Xtandi®, "Xtandi is a trademark of Astellas Pharma, Inc." ) and abiraterone (Zygita®, "Zytiga is a trademark of Janssen Biotech, Inc."). The study will be conducted in two parts. Part 1, a dose escalation phase, will establish RP2D of afuresertib when administered with enzalutamide or abiraterone. Part 2, a dose expansion phase, will further evaluate long-term safety of the combinations at the RP2Ds in additional subjects. Dose-finding cohorts will be studied in parallel and will evaluate safety and pharmacokinetic to guide selection of the dose regimens for further evaluation. Part 2 will begin once the RP2Ds have been established in Part 1. Additional doses and/or schedules may be explored if warranted, based upon the pharmacokinetic (PK) and pharmacodynamic (PD) assessments or emerging preclinical evidence. Overall, approximately 60 chemotherapy-naïve subjects with mCRPC and who are receiving either enzalutamide or abiraterone will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent provided
* Males >=18 years of age (at the time consent is obtained)
* Histologically or cytologically confirmed diagnosis of metastatic prostate adenocarcinoma, without neuroendocrine or small cell features
* Surgically or medically castrated, with testosterone levels of <=50 nanogram (ng)/deciliter (dL) (<=1.73 nanomolar [nM]). If the subject is being treated with luteinizing hormone releasing hormone analogs (subjects who have not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to Cycle 1 Day 1 and must be continued throughout the study.
* Rising Prostate-specific antigen (PSA) after initial response to enzalutamide or abiraterone without radiographic or symptomatic evidence of progression (per Prostate Cancer Working Group 2 criteria): Most recent enzalutamide dose received is 160 milligram (mg) once daily with no change in dose for at least 4 weeks prior to Cycle 1, Day 1. Most recent abiraterone dose received is 1000 mg once daily with prednisone 5 mg twice daily (BID), with no change in dose for at least 2 weeks prior to Cycle 1, Day 1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Able to swallow and retain orally administered medication.
* Adequate baseline organ function defined as: Absolute neutrophils count>=1.5 x 10^9/Liter (L), hemoglobin>=9 grams (g)/dL, Platelets>=75 x 10^9/L, Prothrombin time/International normalized ratio<=1.3 x Upper limit of normal (ULN), Partial thromboplastin time<=1.3 x ULN, Albumin>=2.5 g/dL, Total bilirubin<=1.5 ULN, Aspartate aminotranseferase and Alanine aminotransferase <=2.5 x ULN, Serum creatinine<=ULN OR Estimated glomerular filtration rate>=30 millilite per Minute (mL/min), Fasting Serum Glucose <126 mg/dL, Hemoglobin A1C<=8%. Note: Subjects with ALT or bilirubin values outside the ranges noted in the table above due to Gilbert's syndrome or asymptomatic gallstones are not excluded.
* Male subject with a female partner of childbearing potential must either have a prior vasectomy or agree to use effective contraception from time of first dose of study treatment until 3 months after last dose of study treatment.

Exclusion Criteria:

* Prior treatment with cytotoxic chemotherapy or inhibitors of the Phosphoinositide 3-kinase (PI3K)/protein kinase B (AKT)/ mechanistic target of rapamycin (mTOR) pathway.
* Any investigational drug(s) within 30 days or 5 half-lives of enrollment, whichever is longer.
* Prior malignancy other than Castrate-resistant prostate cancer (CRPC). Exception: Subjects who have been disease-free of the prior malignancy for 3 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Any unresolved >=Grade 2 (per Common Toxicity Criteria for Adverse Events 4.0) toxicity from previous anti-cancer therapy at the time of enrollment, except alopecia or Grade 2 anemia (if hemoglobin is >9.0 gram (g)/dL).
* Presence of any clinically significant gastrointestinal (GI) abnormality or other condition(s) that may alter absorption such as malabsorption syndrome or major resection of the stomach or substantial portion of the small intestine. NOTE: If clarification is needed as to whether a GI abnormality, condition or resection will significantly affect the absorption of study treatment, contact the Sponsor's Medical Monitor.
* Major surgery, radiation therapy, or immunotherapy within 28 days prior to enrollment.
* Known active infection requiring intravenous (IV) or oral anti-infective treatment.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal or cardiac disease).
* For those subjects who will receive afuresertib plus enzalutamide: History of seizures, underlying brain injury with loss of consciousness, transient ischemic attack in the past 12 months, cerebral vascular accident, brain metastases, brain arteriovenous malformation, or use of concomitant medications that may lower the subjects' seizure threshold.
* History or evidence of cardiovascular risk including any of the following:

Clinically significant ECG abnormalities including second degree (Type II) or third degree atrioventricular block.

History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, stenting, or bypass grafting within the past 6 months prior to enrollment.

Class III or IV heart failure as defined by the New York Heart Association functional classification system Left ventricular ejection fraction (LVEF) below 50% Known cardiac metastases Corrected QT interval of >470 millisecond (msec) (or >480 msec with bundle branch block)

* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to afuresertib, enzalutamide, abiraterone, or excipients.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Have a known Human Immunodeficiency Virus (HIV) infection.
* Subjects who are Hepatitis B surface antigen (HbSAg) positive.
* Subjects with a positive test for Hepatitis C virus (HCV) antibody, regardless of viral load. (Note: the subject is eligible if a confirmatory recombinant immunoblot assay [RIBA] test is negative).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), serious adverse events (SAEs) and dose limiting toxicities as a safety measure. | From first dose of study drug until 30 days after last dose of study drug (assessed up to average of 6 months).
  All AEs and SAEs will be collected and recorded from receipt of first dose of study drug until 30 days after the last dose of study drug, or until the start of subsequent therapy.
Change from baseline in composite of laboratory parameters as a safety measure: hematology, clinical chemistry and urinalysis. | From baseline up to end of treatment (assessed up to average of 6 months).
  Changes in the laboratory parameter including hematology, clinical chemistry and urinalysis will be assessed as a measure of safety tolerability and to establish RP2D.
Change from baseline in electrocardiogram values as a safety measure. | From baseline up to average of 6 months.
  Changes in electrocardiograms (ECGs) values will be assessed as a measure of safety, tolerability and to establish RP2D.
Change from baseline in composite of vital signs as a safety measure: blood pressure, temperature and pulse rate. | From baseline up to end of treatment (assessed up to average of 6 months).
  Changes in vital sign values of blood pressure, temperature and pulse rate will be assessed as a measure of safety, tolerability and to establish RP2D.
Composite of PK parameters as a measure of RP2D following administration of afuresertib plus enzalutamide or afuresertib plus abiraterone: AUC and Cmax. | Pre-dose Sample on Day 1 of Cycle 1, 2, 3, 4, and then every 12 weeks and again on Day 1 of Cycle 7 (assessed up to 169 days).
  PK parameters of area under time concentration curve (AUC) and maximum plasma concentration (Cmax) will be evaluated to determine RP2D of afuresertib.
Composite of PK parameters as a measure of RP2D following administration of afuresertib plus abiraterone: AUC and Cmax. | Pre-dose and 2 hours post dose sample will be collected on Day 8 of Cycle 1.
  PK parameters of area under time concentration curve (AUC) and maximum plasma concentration (Cmax) will be evaluated.
Number of participants with adverse events, serious adverse events and dose limiting toxicities to establish RP2D of afuresertib. | Cycle 1 (28 days).
  All AEs and SAEs will be collected and recorded from receipt of first dose of study drug until 30 days after the last dose of study drug, or until the start of subsequent therapy.
Change from baseline in composite of laboratory parameters to establish RP2D of afuresertib: hematology, clinical chemistry and urinalysis. | From baseline up to 28 days (Cycle 1).
  Changes in the laboratory parameter including hematology, clinical chemistry and urinalysis will be assessed as a measure of safety tolerability and to establish RP2D.
Change from baseline in electrocardiogram values to establish RP2D of afuresertib. | From baseline up to 28 days (Cycle 1).
  Changes in electrocardiograms (ECGs) will be assessed as a measure of safety, tolerability and to establish RP2D.
Change from baseline composite of vital sign values to establish RP2D of afuresertib: blood pressure, temperature and pulse rate. | From baseline up to 28 days (Cycle 1).
  Changes in vital sign values of blood pressure, temperature and pulse rate will be assessed as a measure of safety, tolerability and to establish RP2D.

SECONDARY OUTCOMES:
Composite of afuresertib PK parameters following administration with enzalutamide: AUC and Cmax. | Blood samples will be collected at pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post dose on Day 1of Cycle 1.
  PK profile of afuresertib will be established following administration with enzalutamide by assessing AUC and Cmax.
Composite of enzalutamide PK parameters following administration alone and in combination with afuresertib: AUC and Cmax. | Blood samples will be collected at pre-dose, 0.5, 1, 2, 3, 4, 6 and 24 hours post dose on Day-1 and Day 1 in Cycle 2.
  PK profile of enzalutamide will be establish by assessing AUC and Cmax when administered alone and in combination with afuresertib.
Composite of PK parameters following administration afuresertib and abiraterone alone and in combination with each other: AUC and Cmax. | Blood samples will be collected at pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post dose on Day 15 of Cycle 1 and Day 1 of Cycle 2 for afuresertib and on Day-1 and Day 1 in Cycle 2 for abiraterone.
  PK profile of afuresertib and abiraterone will be establish by assessing AUC and Cmax when administered alone and in combination with each other.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline